CLINICAL TRIAL: NCT06279156
Title: Optimal Frequency of Total Body Water Measurements by Bioelectrical Impedance Analysis to Prevent Intradialytic Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University Hospital (Other)
Responsible Party: Principal Investigator, Aphichat Chatkrailert, Thammasat University Hospital, Thammasat University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MTU-EC-IM-0-014/65
Record Dates: First submitted 2024-02-18; First posted 2024-02-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Intradialytic Hypotension; End Stage Renal Disease on Dialysis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the first group (every-1-month BIA and then every-2-month BIA) (Experimental): measure Bioelectrical Impedance analysis (BIA) for patients' dry weight every 1 month for 4 months, and then every 2 months for 4 months
  Interventions: Device: Bioelectrical Impedance Analysis (BIA)
- the second group (every-2-month BIA and then every-1-month BIA) (Experimental): measure Bioelectrical Impedance analysis (BIA) for patients' dry weight every 2 months for 4 months, and then every 1 month for 4 months
  Interventions: Device: Bioelectrical Impedance Analysis (BIA)

INTERVENTIONS:
Device: Bioelectrical Impedance Analysis (BIA) — Measure BIA for patients' dry weight to compare between measuring every-1-month or every-2-month.
  In brief, BIA is the machine used for measure body components such as fat, muscle, and free water. It relies on the principle of using the multifrequency of low electric currents to the body and measurement of the ability of the electrical currents passing different body composition. Thus, the machine can calculate back for the amount of each body composition.

SUMMARY:
The goal of this clinical trial was to compare the efficiencies of bioelectrical impedance analysis (BIA) measurement frequency in preventing intradialytic hypotension in end-stage renal disease (ESRD) patients undergoing regular hemodialysis. The main question aimed to answer about the optimum frequency of BIA measurements to prevent intradialytic hypotension.

Participants underwent BIA measurements to determine their appropriate dry weight, and factors affecting intradialytic hypotension.

Researchers compared the efficiencies of BIA measurements between the every-1-month group and the every-2-month group to prevent intradialytic hypotension.

DETAILED DESCRIPTION:
The study, conducted at Thammasat University Hospital, aimed to assess the efficacy of different frequencies of BIA measurements in preventing intradialytic hypotension in ESRD patients undergoing hemodialysis.

The trial enrolled ESRD patients and collected data from June 2022 to February 2023.

Research Procedure:

* Screening for eligibility was conducted among individuals undergoing hemodialysis at the hemodialysis unit of Thammasat University Hospital.
* Informed consent was obtained from participants or their authorized representatives.
* Basic demographic and medical data were recorded, including gender, age, pre-existing conditions, causes of kidney disease, smoking habits, regular medications. The dry weight, interdialytic weight gain (IDWG), and net ultrafiltration (UF) were calculated from every session of the patient's dialysis, and then taken the average. Blood flow rate (BFR) and dialysate temperature were taken from the largest value from each dialysis session and the greatest frequency. Single pool KT/V and blood tests (hemoglobin, serum albumin, electrolytes) were from the closest value before entering the research. Pre-dialysis systolic blood pressure (SBP) and diastolic blood pressure (DBP) were the average values.
* Volunteers were randomly assigned to two groups, each consisting of 45 individuals. Group 1 underwent BIA measurements monthly for 4 months, then switched to bi-monthly BIA measurements for 4 months. Group 2 underwent BIA measurements every 2 months for 4 months, then switched to monthly BIA measurements for 4 months. Data were used as a combination to adjust dry weight for accurate fluid removal.
* Episodes of intra-dialyltic hypotension were recorded and the numbers of such episodes were calculated as incidence rates to explore the most optimum frequency of BIA measurement (between every-1-month group and the every-2-month). Intradialytic hypotension in this study was defined as a decrease in (SBP) ≥ 20 mmHg or a decrease in mean arterial pressure (MAP) ≥ 10 mmHg. For BIA measurements in addition to the presence of intradialytic hypotension, the number of occurrences of intradialytic hypotension was counted as one increase.
* Factors affecting intradialytic hypotension were also explored.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* dialysis vintage ≥ 3 months
* hemodialysis at least thrice weekly
* hemodialysis ≥ 3 hours per session.

Exclusion Criteria:

* congestive heart failure (NYHA class 3-4)
* cardiac arrhythmias with relapse within 1 month and still unable to control symptoms during the drug adjustment period
* coronary artery disease which active within 1 month without treatment
* patients who take regular oral medications to raise blood pressure before undergoing dialysis such as midodrine
* patients with low blood pressure or requiring blood pressure medication adjustments within 1 month period
* has another unstable symptom

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
incidence rate ratio of intra-dialytic hypotension of every-1-month BIA to every-2-month BIA | In each 4-month period of each assigned intervention group during hemodialysis sessions (48 hemodialytic sessions of each patient in each group), or total observation time was 8 months (96 hemodialytic sessions of each patient in both groups).
  Numbers of intra-dialytic hypotension sessions which each patient experiences when apply every-1-month BIA or every-2-month BIA will be collected. Then, the incidence rate of intra-dialytic hypotension (numbers of intra-dialytic hypotension episodes/numbers of total hemodialytic episodes) of every-1-month BIA or every-2-month BIA will be calculated. Finally, incidence rate ratio of intra-dialytic hypotension of every-1-month BIA to every-2-month BIA will be calculated.

SECONDARY OUTCOMES:
factors affecting intra-dialytic hypotension | In each 4-month period of each assigned intervention group (every-1-month BIA, and every-2-month BIA) during hemodialysis sessions (total observation time was 8 months).
  The incidence rate ratio (numbers of intra-dialytic hypotension episodes/numbers of total hemodialytic episodes) will be calculated to explore whether individual parameters; for example, sex, age, underlying diseases, type of medication uses, data prior or during hemodialysis ( e.g. dialysis-vintage year, blood flow rate, interdialytic weight gain, etc.) or laboratory data relate to incidence rate ratio of intradialytic hypotension, or not.

CONTACTS AND LOCATIONS:
Overall Officials: Aphichat Chatkrailert, M.D., Principal Investigator — Thammasat University Hospital
Locations (1):
- Thammasat University Hospital, Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: No
There was no plan to share IPD to other researchers. We used IPD in internal work only.

REFERENCES:
- [Result] Zhang M, Wang M, Li H, Yu P, Yuan L, Hao C, Chen J, Kalantar-Zadeh K. Association of initial twice-weekly hemodialysis treatment with preservation of residual kidney function in ESRD patients. Am J Nephrol. 2014;40(2):140-50. doi: 10.1159/000365819. Epub 2014 Aug 23. PMID 25171342
- [Result] Agarwal R, Alborzi P, Satyan S, Light RP. Dry-weight reduction in hypertensive hemodialysis patients (DRIP): a randomized, controlled trial. Hypertension. 2009 Mar;53(3):500-7. doi: 10.1161/HYPERTENSIONAHA.108.125674. Epub 2009 Jan 19. PMID 19153263
- [Result] Breidthardt T, McIntyre CW. Dialysis-induced myocardial stunning: the other side of the cardiorenal syndrome. Rev Cardiovasc Med. 2011;12(1):13-20. doi: 10.3909/ricm0585. PMID 21546884
- [Result] Lee Y, Okuda Y, Sy J, Kim SR, Obi Y, Kovesdy CP, Rhee CM, Streja E, Kalantar-Zadeh K. Ultrafiltration Rate Effects Declines in Residual Kidney Function in Hemodialysis Patients. Am J Nephrol. 2019;50(6):481-488. doi: 10.1159/000503918. Epub 2019 Oct 29. PMID 31661683
- [Result] Kanbay M, Ertuglu LA, Afsar B, Ozdogan E, Siriopol D, Covic A, Basile C, Ortiz A. An update review of intradialytic hypotension: concept, risk factors, clinical implications and management. Clin Kidney J. 2020 Jul 8;13(6):981-993. doi: 10.1093/ckj/sfaa078. eCollection 2020 Dec. PMID 33391741
- [Result] Kim HR, Bae HJ, Jeon JW, Ham YR, Na KR, Lee KW, Hyon YK, Choi DE. A novel approach to dry weight adjustments for dialysis patients using machine learning. PLoS One. 2021 Apr 23;16(4):e0250467. doi: 10.1371/journal.pone.0250467. eCollection 2021. PMID 33891656
- [Result] Kyle UG, Bosaeus I, De Lorenzo AD, Deurenberg P, Elia M, Gomez JM, Heitmann BL, Kent-Smith L, Melchior JC, Pirlich M, Scharfetter H, Schols AM, Pichard C; Composition of the ESPEN Working Group. Bioelectrical impedance analysis--part I: review of principles and methods. Clin Nutr. 2004 Oct;23(5):1226-43. doi: 10.1016/j.clnu.2004.06.004. PMID 15380917
- [Result] Brunani A, Perna S, Soranna D, Rondanelli M, Zambon A, Bertoli S, Vinci C, Capodaglio P, Lukaski H, Cancello R. Body composition assessment using bioelectrical impedance analysis (BIA) in a wide cohort of patients affected with mild to severe obesity. Clin Nutr. 2021 Jun;40(6):3973-3981. doi: 10.1016/j.clnu.2021.04.033. Epub 2021 Apr 28. PMID 34139470